CLINICAL TRIAL: NCT04559412
Title: Phase 1b Proof-of-concept, Open-label Study to Assess the Safety and Pilot Efficacy of Enbrel® Administered by the Sofusa® DoseConnect™ Delivery System for the Treatment of Rheumatoid Arthritis
Brief Title: Study to Assess the Safety and Efficacy of Enbrel Administered by Sofusa DoseConnect for Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STI-SOFUSA-1003
Record Dates: First submitted 2020-09-03; First posted 2020-09-22 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sofusa Enbrel (Experimental): Enbrel® administered by the Sofusa® DoseConnect™ delivery system
  Interventions: Device: Sofusa DoseConnect; Drug: Enbrel

INTERVENTIONS:
Device: Sofusa DoseConnect — 25 to 50 mg Enbrel® administered by the Sofusa® DoseConnect™ delivery system once weekly for 12 weeks
  Other Names: sofusa
Drug: Enbrel — 25 to 50 mg Enbrel® administered by the Sofusa® DoseConnect™ delivery system once weekly for 12 weeks

SUMMARY:
This is an open-label pilot study in patients with rheumatoid arthritis (RA). All patients will receive SOFUSA Enbrel 25 mg once weekly. The dose will be increased to 50 mg if the dose escalation criteria are met during the dose escalation phase of the study.

DETAILED DESCRIPTION:
This study is a Phase 1b proof-of-concept, open-label study to assess the safety and pilot efficacy of Enbrel administered by the Sofusa® DoseConnect™ delivery system (SOFUSA) for the treatment of patients with moderately to severe RA and an inadequate response to subcutaneous (SC) Enbrel. SOFUSA Enbrel will be administered once weekly to patients for 12 weeks. Patients will start on an Enbrel dose of 25 mg during the induction phase of the study and may be increased to an Enbrel dose of 50 mg during the dose escalation phase of the study based on the dose escalation criteria. Patients will remain on either the 25 mg or 50 mg dose for the final maintenance phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Has rheumatoid arthritis (RA) as defined by having a score of 6 or higher on the 2010 ACR-EULAR classification criteria
* Is currently on Enbrel therapy and has received once-weekly Enbrel injections for at least 12 weeks with no more than 1 missed dose in the 12 weeks prior to Screening.
* Must meet the following disease criteria:

Have a DAS28(CRP) score > 2.9 at Screening Have a DAS28(ESR) score > 3.2 at Screening Swollen joint count ≥ 3 (28-joint count) and Tender joint count ≥ 3 (28-joint count) at Screening and Baseline

* If on oral or subcutaneous MTX (up to 25 mg/week) or other permitted oral conventional synthetic disease-modifying anti-rheumatic drugs (DMARDs) (i.e., leflunomide, up to 20 mg/day; hydroxychloroquine, up to 400 mg/day; or sulfasalazine, up to 3 g/day), must be on stable dose (MTX ≥ 12 weeks and other permitted DMARDs ≥ 8 weeks) within the specified ranges prior to Baseline. Note: if on methotrexate (MTX), subjects must be on a stable dose of folic acid (total ≥ 5 mg per week for ≥ 12 weeks) prior to Baseline and must continue a stable dose during the course of the study.
* If taking regular nonsteroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase-2 (COX-2) inhibitors, paracetamol/acetaminophen, or oral glucocorticoids for treatment of RA symptoms, must be on stable dose and route of administration for at least 2 weeks before Baseline
* Females of childbearing potential must agree to use acceptable method(s) of contraception for the duration of the study and for 3 months after the last dose of study drug

Exclusion Criteria:

* Has participated in a clinical trial with a drug or device within 30 days prior to Screening
* Prior treatment with investigational therapy within 30 days or 5 half-lives before Screening (whichever is longer)
* History of hypersensitivity to any recombinant protein drugs or any of the excipients used in Enbrel
* Has skin contact sensitivities (due to SOFUSA device adhesive) or allergies to iodine (due to the iodine in ICG)
* Lack of any clinical response to Enbrel in the Investigator's opinion
* Treatment with other biologic agents (e.g., interleukin [IL] 6, IL17, IL12/23 inhibitors; abatacept, tumor necrosis factor [TNF] inhibitors) besides Enbrel within 24 weeks before Baseline
* Previous treatment with more than 2 other tumor necrosis factor (TNF) inhibitor therapies (besides Enbrel), more than 2 targeted therapies with different mechanisms of action (e.g., Janus kinase inhibitors, T cell costimulation inhibitor, IL-6 receptor antagonist), or any cell depleting agents (e.g., anti-CD20)
* Use of chlorambucil or cyclophosphamide within 24 weeks of Baseline
* Use of leflunomide within 8 weeks of Baseline, if washing out of leflunomide, unless a cholestyramine washout has been performed, then use of leflunomide within 4 weeks of Baseline
* Use of MTX, hydroxychloroquine, or sulfasalazine within 4 weeks of Baseline, if washing out of MTX, hydroxychloroquine, or sulfasalazine
* Any systemic nonbiologic DMARD (e.g., Janus kinase inhibitor, cyclosporine, azathioprine) within 4 weeks of Baseline
* History of or ongoing inflammatory, autoimmune, or painful musculoskeletal diseases (except for Sjogren's syndrome or fibromyalgia) which could interfere with the RA assessments as determined by the Investigator
* Functional RA status of class IV according to the ACR 1991 revised criteria at Screening or Baseline
* Oral glucocorticoids > 10 mg/day prednisone equivalent within 4 weeks prior to Baseline
* Opioid tolerant: defined as the use of opiate analgesics at a dose of > 30 mg/day of oral morphine equivalent on 4 of the last 7 days prior to Baseline
* Use of intramuscular, intravenous, or intraarticular corticosteroid therapy within 4 weeks prior to Baseline
* Treatment with any intra-articular hyaluronic acid preparation within 12 weeks prior to Baseline
* Chronic arthritis diagnosis before the age of 17 years
* Presence of any extra-articular manifestations of RA, except for rheumatoid nodules
* Joint surgery within the preceding 8 weeks before Screening
* History of, or presence of cancer (if < 5 years from successful treatment even with no evidence of recurrent disease) or lymphoproliferative or hematologic disease, other than a successfully and completely treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix and/or removed non-invasive colon or bladder polyps, with no evidence of recurrence
* History of uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (New York Heart Association III-IV), active peptic ulcer disease, recent stroke, myocardial infarction, or thromboembolism (within 6 months), or any other condition which, in the opinion of the Investigator, would put the patient at risk by participation in the study
* Previous diagnosis or signs of demyelinating disease
* History of clinically significant hematologic (e.g. severe anemia, leukopenia, thrombocytopenia), renal or liver disease (e.g. glomerulonephritis, fibrosis, cirrhosis, hepatitis) or abnormal clinical laboratory tests at Screening
* Receipt of any blood products within 12 weeks of Baseline
* History of persistent chronic infection; recurrent infection (more than 3 infections requiring antimicrobial therapy within the last 12 months); or active infections requiring hospitalization or treatment with systemic anti-infective therapy within 4 weeks before Screening (counted from anti-infective therapy stop date), except for fungal infection of nails or nail beds
* History of or current active tuberculosis or presence of latent tuberculosis as detected by imaging (e.g., chest radiograph) and/ or QuantiFERON®-TB Gold Plus test (QFT) NOTE: Positive QFT (or 2 or more tests that are indeterminate) and/or positive imaging result (within 12 weeks prior to Screening or at Screening) excludes a patient from participation in the study (except for patients who have documentation of completing an acceptable regimen for treatment of latent tuberculosis with no known re-exposure to tuberculosis since treatment completion)
* History or evidence of opportunistic infections (eg, histoplasmosis, listeriosis, legionellosis)
* Known immune deficiency, known human immunodeficiency virus (HIV) positive or positive at Screening, or immunocompromised for other reasons
* Serology positive for hepatitis B virus (HBV) surface antigen (HBsAg) or core antibody (HBcAb) or hepatitis C virus (HCV) antibody (HCV-Ab) or ribonucleic acid (HCV RNA). Patients treated for HCV and considered cured (negative HCV RNA) may participate in the study
* Positive RT-PCR or the equivalent COVID-19 test at Screening
* History or evidence of ongoing significant drug or alcohol abuse
* Known depression or other psychiatric condition, which in the Investigator's opinion may decrease likelihood of participant adherence to the study protocol requirements
* History of vaccination with live vaccines within the preceding 8 weeks prior to Baseline or known to require vaccination with live vaccines during the study period
* For female participants, currently breastfeeding (lactating) or less than 12 weeks from cessation of lactation
* Pregnant woman where pregnancy is defined as the state of a woman after conception and until the termination of gestation, confirmed by a positive serum pregnancy test at Screening or positive urine pregnancy test at Baseline
* Patient is considered by the Investigator, for any reason, to be an unsuitable candidate for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and their relationships to SOFUSA administration | Baseline through Week 12
  Incidence and severity of adverse events and their relationships to SOFUSA administration

SECONDARY OUTCOMES:
Change in Disease Activity Score 28-joint count C reactive protein (DAS28(CRP)) | Baseline to Week 12
  Change from Baseline in DAS28(CRP) score at Week 12
Change in DAS28(CRP) score over time | Baseline through Week 12
  Change from Baseline in DAS28(CRP) score over time
Change in Disease Activity Score 28-joint count erythrocyte sedimentation rate (DAS28(ESR)) over time | Baseline through Week 12
  Change from Baseline in DAS28(ESR) score over time
Change in Simplified Disease Activity Index (SDAI) score over time | Baseline through Week 12
  Change from Baseline in SDAI score over time
Change in Clinical Disease Activity Index (CDAI) score over time | Baseline through Week 12
  Change from Baseline in CDAI score over time
Proportion of patients with low disease activity (LDA) over time as assessed by the DAS28(CRP) | Baseline through Week 12
  Proportion of patients with DAS28(CRP) score < 2.9 over time
Proportion of patients with LDA over time as assessed by the DAS28(ESR) | Baseline through Week 12
  Proportion of patients with DAS28(ESR) score ≤ 3.2 over time
Proportion of patients with LDA over time as assessed by the SDAI | Baseline through Week 12
  Proportion of patients with SDAI score ≤ 11.0 over time
Proportion of patients with LDA over time as assessed by the CDAI | Baseline through Week 12
  Proportion of patients with CDAI score ≤ 10 over time
Proportion of patients achieving ACR20/50/70 response over time | Baseline through Week 12
  Proportion of patients achieving ACR20/50/70 response over time
Proportion of patients achieving moderate or good EULAR response over time | Baseline through Week 12
  Proportion of patients achieving moderate or good EULAR response over time
Proportion of patients achieving a minimally clinically important difference (MCID) of 0.22 in the Health Assessment Questionnaire-Disability Index (HAQ-DI) over time | Baseline through Week 12
  Proportion of patients achieving a MCID of 0.22 in HAQ-DI over time

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD JD MBA, Study Director — Sorrento Therapeutics
Locations (1):
- Atlanta Research Center for Rheumatology, Atlanta, Georgia, United States